CLINICAL TRIAL: NCT05202795
Title: Provider Perspectives on the Postpartum Pain Experience and Attitudes About Pain Management
Brief Title: Postpartum Pain Experience and Attitudes About Opioid Prescribing
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Nevert Badreldin, Assistant Professor of Obstetrics and Gynecology (Maternal Fetal Medicine), Northwestern University
Other Study IDs: STU00215779
Record Dates: First submitted 2022-01-05; First posted 2022-01-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Postpartum Pain; Pain Management; Opioid Prescribing
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective qualitative study of obstetric clinicians examining factors which influence their approach to postpartum pain management, their perspectives and preferences of interventions aimed at reducing opioid use, and the biases which may contribute disparities in this setting.

DETAILED DESCRIPTION:
Opioid misuse has been declared a national emergency in the United States. More than half of hospitalized patients receive an opioid during their hospitalization. As birth is the most common reason for hospitalization, reproductive-aged individuals are particularly vulnerable to opioid exposure and are an important population for addressing the opioid epidemic. Indeed, data have demonstrated the high frequency of postpartum inpatient and outpatient opioid use, the wide variation in postpartum pain management, the lack of alignment of opioid prescribing with patient reports of pain, and the contributions of obstetric clinicians to opioid prescribing.

The opioid epidemic has a differential impact by race/ethnicity; individuals of minority race/ethnicity are less likely to receive an opioid for pain management than non-Hispanic White individuals. Notably, data show that, despite reporting higher levels of pain postpartum, minority race/ethnicity birthing individuals receive less opioid treatment as inpatients and are less frequently prescribed an opioid upon hospital discharge. A complete understanding and, ultimately improvement, of these experiences and reduction in disparities requires a deeper delve into influences which guide clinicians in their management of postpartum pain.

This investigation aims to fill an unmet need for a systematic, in-depth, and unbiased evaluation of obstetric clinicians' experience of postpartum pain management. This is a prospective qualitative study of obstetric clinicians, examining factors which influence their approach to postpartum pain management, biases which may contribute to disparities, and their perspectives and preferences of interventions to reduce opioids and improve pain control. Investigators will conduct in-depth semi-structured interviews with up to 50 obstetric clinicians, including physicians, advanced practitioners, and nurses. Aim 1 will evaluate beliefs and factors which influence clinicians' management of postpartum pain, including potential clinician-level biases which may contribute to disparities. Using the Consolidated Framework for Implementation Science, Aim 2 will evaluate clinicians' perspectives and preferences of interventions to reducing postpartum opioid prescribing and improving pain control, in order to optimize the implementation of future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Practicing health care provider in obstetrics/gynecology at Northwestern Medicine

Exclusion Criteria:

* Below the age of 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Practicing health care providers in obstetrics/gynecology
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Factors which influence clinicians' management of postpartum pain | through study completion, an average of 1 year
  Through analysis of qualitative interviews, themes such as approaches to pain management, awareness of disparities in pain management, and beliefs about cultural and social influences of pain will be reviewed. The constant comparative method will be applied.

SECONDARY OUTCOMES:
Clinicians' perspectives and preferences for interventions targeted at reducing postpartum opioid prescribing | through study completion, an average of 1 year
  Through analysis of qualitative interviews, themes such as knowledge, acceptability, barriers, feasibility, health impact, and perceived need will be reviewed for different types of interventions to reduce opioid prescribing.

CONTACTS AND LOCATIONS:
Overall Officials: Nevert Badreldin, MD, MS, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No